CLINICAL TRIAL: NCT06261359
Title: A Phase II, Randomized, Double-blind, Multi-center, Placebo-Controlled Study of the Efficacy and Safety of CEND-1 in Combination With Chemotherapy as First-Line Therapy in Patients With Locally Advanced Unresectable or Metastatic Pancreatic Ductal Adenocarcinoma
Brief Title: A Study of CEND-1 With Chemotherapy as First-Line Therapy in Patients With Pancreatic Ductal Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CEND1-202
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2023-11

CONDITIONS: Pancreatic Ductal Adenocarcinoma (PDAC)
MeSH Terms: interventions — Gemcitabine; Taxes; Albumin-Bound Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CEND-1+ nab-paclitaxel + gemcitabine (Experimental): Participants will receive nab-paclitaxel 125mg/m2; CEND1 3.2mg/kg IV; and then Gemcitabine 1000mg/m2, on Day 1, 8 and 15 of each cycle. Each cycle will be 28 days.
  Interventions: Drug: CEND-1; Drug: Gemcitabine; Drug: Nab paclitaxel
- Placebo+ nab-paclitaxel + gemcitabine (Placebo Comparator): Participants will receive nab-paclitaxel 125mg/m2; placebo IV; and then Gemcitabine 1000mg/m2, on Day 1, 8 and 15 of each cycle. Each cycle will be 28 days.
  Interventions: Drug: Gemcitabine; Drug: Nab paclitaxel

INTERVENTIONS:
Drug: CEND-1 — CEND-1 will be provided as concentrate for solution to be administered via IV injection.
  Other Names: iRGD; LSTA1; certepetide
  Arms: CEND-1+ nab-paclitaxel + gemcitabine
Drug: Gemcitabine — Gemcitabine will be provided as solution to be administered via IV infusion.
  Other Names: Gemzar
Drug: Nab paclitaxel — Nab-paclitaxel will be provided as solution to be administered via IV infusion.
  Other Names: Abraxane

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of CEND-1 in combination with gemcitabine/nab-paclitaxel versus gemcitabine/nab-paclitaxel and placebo as first-line treatment in patients with Locally Advanced Unresectable or Metastatic Pancreatic Ductal Adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* 18~80 years old, male or female;
* Locally advanced unresectable or metastatic PDAC confirmed by histopathology or cytopathology;
* Patients who have not received prior systemic therapy for locally advanced or metastatic pancreatic cancer;
* Patients with at least one measurable tumor lesion per RECIST v1.1;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* Expected survival time ≥ 12 weeks;
* Patients who have adequate organ function;
* Female subjects who are not pregnant or not breastfeeding. A negative pregnancy test for females of childbearing potential within 7 days prior to first dosing. Male and female subjects of childbearing potential must agree to use highly effective method of contraception during the entire course of the study and within 180 days after the end of the study.
* Subjects participate voluntarily and sign informed consent.

Exclusion Criteria:

* Concurrent use of other anticancer drugs, including chemotherapy, targeted therapy, immunotherapy, or biologics;
* The patients who are known to be allergic to the investigatinal drug or its any excipient;
* Patients with the following conditions: myocardial infarction, severe/unstable angina, NYHA grade 2 or above cardiac dysfunction, and clinically significant supraventricular or ventricular arrhythmia requiring clinical intervention within 6 months before signing the ICF;
* Patients with high risk for gastrointestinal bleeding or abdominal bleeding as assessed by the investigator, such as tumor invasion of the gastro duodenum finger intestines, large blood vessels, etc.;
* Patients with symptomatic CNS metastasis, leptomeningeal metastasis, or spinal cord compression due to metastasis.
* Patients with other active malignant tumors within 3 years before signing the ICF. Patients with cured skin basal cell carcinoma or squamous cell carcinoma, carcinoma in situ of the cervix, carcinoma in situ of the breast ductal, and papillary thyroid cancer can be enrolled.
* Patients with human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), active hepatitis or co-infection with hepatitis B and C.
* Patients who require systemic antibiotics for ≥7 days within 4 weeks prior to first dose, or unexplained fever >38.5°C prior during screening or before first dose;
* Patients who participated in any other clinical studies;
* Patients with a known history of psychoactive drug abuse, alcohol abuse, or substance abuse; History of definitive neurological or mental disorder, including epilepsy or dementia;
* The patients with added risks associated with the study or may interfere with the interpretation of study results as determined by the investigator, or deemed unsuitable by the investigator and/or sponsor.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-03-19 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Approximately 36 months
  ORR is defined as the proportion of participants who have a best overall response of Complete Response (CR) or Partial Response (PR) as assessed by investigator evaluation per RECIST 1.1.

SECONDARY OUTCOMES:
Overall Survival (OS) | Approximately 36 months
  OS is defined as the duration from randomization to the time point when death occurs due to any cause.
Progression Free Survival(PFS) | Approximately 36 months
  PFS is defined as the duration from randomization to the first imaging confirmation of progressive disease per RECIST 1.1 by investigator evaluation or death due to any cause (whichever occurs first).
6-month PFS rate | Approximately 36 months
  6-month progression-free survival (PFS) rate.
Duration Of Response (DOR) | Approximately 36 months
  DOR is defined as the time from the date of the first response (CR/PR) until the date of progressive disease as assessed by investigator evaluation per RECIST 1.1 or death due to any cause (whichever occurs first).
Disease Control Rate (DCR) | Approximately 36 months
  DCR was defined as the percentage of confirmed CR, PR or stable disease at the best response as assessed by investigator evaluation per RECIST 1.1.
Incidence of AEs, SAEs and treatment-emergent adverse events (TEAEs) | From the subject signs the ICF to 30 days after the last dose of study drug was administered.
  Adverse events (AEs), serious adverse events (SAEs), treatment-emergent adverse events are included. The investigator should carry out judgment for investigational drug correlation.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese People's Liberation Army (PLA) General Hospital, Beijing, Beijing Municipality, China